CLINICAL TRIAL: NCT05972876
Title: MRI-based Graft Maturity After Blood Flow Restriction Training in Bone-patellar Tendon-bone Anterior Cruciate Ligament Reconstruction: a Randomized Controlled Study
Brief Title: Graft Maturity After Blood Flow Restriction Training in ACL Reconstruction
Acronym: TimeToMature
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL83376.096.22
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Bone-Patellar Tendon-Bone Grafting
Keywords: Blood Flow Restriction Therapy
MeSH Terms: interventions — Blood Flow Restriction Therapy; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood flow restriction training (BFRT) (Experimental): Patients in the BFRT group will perform four sets (30, 15, 15 and 15 repetitions, respectively) of unilateral leg press, seated leg extension, deadlift and squat exercises with 30s inter-set rest periods throughout a 0-90° range of motion at 30% one-repetition maximum
  Interventions: Behavioral: Blood flow restriction training
- Resistance training (RT) (Active Comparator): Patients in the resistance training group will perform 3x10 reps (30s inter-set rest) of unilateral leg press, seated leg extension, deadlift and squat exercises exercise throughout a 0-90° range of motion with incremental increase in external-load up to 70% of patients' one-repetition maximum
  Interventions: Behavioral: Resistance training

INTERVENTIONS:
Behavioral: Blood flow restriction training — BFR will be achieved using an automatic personalized tourniquet system (MAD-UP, Angers, France) designed to automatically calculate limb occlusion pressure
  Arms: Blood flow restriction training (BFRT)
Behavioral: Resistance training — Resistance training will be performed without any blood flow restriction
  Arms: Resistance training (RT)

SUMMARY:
Rationale Graft maturity is correlated with strength and biomechanical properties of the reconstructed ACL. There are concerns that heavy-load resistance training (HLRT) may have detrimental effects on ACL graft maturation. Therefore, low-load blood flow restriction training (LL-BFRT) has been suggested as an alternative to HLRT. As LL-BFRT is an increasingly popular method for the rehabilitation after an ACL reconstruction, it is important to evaluate the value of this treatment.

Objectives The main objective is to evaluate the effect of LL-BFRT on MRI-based graft maturity after ACL reconstruction compared to HLRT. The secondary objectives are the effect of LL-BFRT on donor-site morbidity, range of motion, knee stability, patient reported outcome measurements, muscle strength, safe return to pre-injury level of sport and patient satisfaction. Furthermore, feasibility and safety of rehabilitation will be assessed.

Study design Randomized controlled trial . Study population Patients who will undergo primary bone-patellar tendon-bone ACL reconstruction and rehabilitation at Knie-Heup centrum Plus will be assessed for eligibility. The exclusion criteria are: venous thromboembolism, sickle cell anemia, severe hypertension, contra-indication for accelerated rehabilitation, contra-indication for MRI scan or patients who are not willing/able to participate.

Intervention LL-BFRT includes 12 weeks of biweekly strength training and starts two weeks after surgery.

Comparison HLRT includes 12 weeks of biweekly strength training and starts two weeks after surgery.

Main study endpoints The main endpoints are MRI-based graft maturity defined as signal-to-noise quotient three and nine months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients (18-64 years) who will undergo primary BPTB reconstruction at Zuyderland Medical Center and rehabilitation at Knie-Heup centrum Plus.

Exclusion Criteria:

* venous thromboembolism, sickle cell anemia, severe hypertension, contra-indication for accelerated rehabilitation, contra-indication for MRI scan or not willing/able to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Graft Maturity | 3 and 9 months after surgery
  Graft maturity will me measured as signal intensity of ACL graft using sagittal proton density-weighted images (PDWI)

SECONDARY OUTCOMES:
Range of motion | 3 and 9 months after surgery
  Range of motion will be evaluated with the use of a goniometer.
Knee stability | 3 and 9 months after surgery
  With patients lying supine in 30° of flexion anterior tibial translation in mm will be measured with the use of a Rolimeter
Anterior knee pain | 3 and 9 months after surgery
  anterior knee pain is measured on the Numeric Rating Scale, 0=no pain and 10=maximum pain
Knee pain and function | 3 and 9 months after surgery
  Knee Osteoarthritis Outcome Score (0 to 100, 0 being the best outcome)
Knee function | 3 and 9 months after surgery
  knee function (measured using the International Knee Documentation Committee, 0 to 100, 100 being the best outcome
patient confidence | 3 and 9 months after surgery
  using the Anterior Cruciate Ligament Return To Sport after Injury scale, 0 to 100, 100 being the best outcome
hamstring strength | 3 and 9 months after surgery
  Patients hamstring (standing leg curl) strength will be measured on the KINEO LEG PRO
isokinetic quadriceps strength | 3 and 9 months after surgery
  Patients isokinetic quadriceps (seated leg extension) will be measured on the KINEO LEG PRO
Return to pre-injury level of sport | 9 months after surgery
  Return to pre-injury level of sport and timing of return to sport will be evaluated by self-report

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Most, Principal Investigator — Zuyderland Medisch Centrum; Baris Koc, MD, PhDc, Study Director — Zuyderland Medisch Centrum
Locations (1):
- Zuyderland Medical Center, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared upon reasonable written request